CLINICAL TRIAL: NCT04382547
Title: Treatment of Covid-19 Associated Pneumonia With Allogenic Pooled Olfactory Mucosa-derived Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC2(Covid)
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: COVID; Covid-19; Coronavirus; Pneumonia; Pneumonia, Viral; Pneumonia, Interstitial; Sars-CoV2
Keywords: pneumonia; Sars-COV2; Covid-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia; Pneumonia, Viral; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): Patients with Covid-19 associated pneumonia receiving standard treatment and allogenic pooled olfactory mucosa-derived mesenchymal stem cells
  Interventions: Biological: Allogenic pooled olfactory mucosa-derived mesenchymal stem cells; Other: Standard treatment according to the Clinical protocols
- control (Active Comparator): Patients with Covid-19 associated pneumonia receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Allogenic pooled olfactory mucosa-derived mesenchymal stem cells — Allogenic pooled olfactory mucosa-derived mesenchymal stem cells
  Arms: mesenchymal stem cells
Other: Standard treatment according to the Clinical protocols — Standard treatment according to the Clinical protocols

SUMMARY:
Treatment of patients with Covid-19 associated pneumonia using intravenous injection of allogenic pooled olfactory mucosa-derived mesenchymal stem cells

DETAILED DESCRIPTION:
During the implementation of the project, it is planned to develop a method for the treatment of severe covid-19 associated interstitial pneumonia using allogeneic mesenchymal stem cells. The positive outlook for the effectiveness of MSCs is due to the following:

* knowledge of the leading role of immunopathogenetic mechanisms in the development of acute interstitial lung diseases and the pronounced immunomodulating properties of MSCs;
* high tropism of MSCs to lung tissue when administered intravenously;
* the ability of MSCs to stimulate tissue regeneration and the effective use of MSCs in the treatment of acute damage to the myocardium and kidneys, which will contribute to the treatment of multiple organ failure;
* positive results of preclinical studies of the method of treatment of viral pneumonia in animals, and the first clinical studies in patients.

ELIGIBILITY:
Inclusion Criteria:

* PCR-confirmed Covid-19 pneumonia
* respiratory failure

Exclusion Criteria:

* diagnosed cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 3 weeks
  Number of patients cured, assessed by PCR in addition to chest CT scan

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events | 3 weeks
  MSC infusion related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Y Hancharou, Dr., Study Director — Director, the Institute of Biophysics and Cell Engineering of NAS of Belarus; Eduard A Dotsenko, Dr., prof., Study Director — Head of the chair, Belarusian State Medical University; Natalia G Antonevich, Dr., Principal Investigator — Head of the Lab of Institute of Biophysics and Cell Engineering of NAS
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No